CLINICAL TRIAL: NCT05100199
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Parallel-Group Phase 2 Study Evaluating the Safety and Efficacy of OnabotulinumtoxinA X for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: A Study to the Assess the Change in Condition and Adverse Events of OnabotulinumtoxinA X Injection in Adult Participants With Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2042-201-008
Record Dates: First submitted 2021-09-30; First posted 2021-10-29 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Glabellar Lines
Keywords: OnabotulinumtoxinA X; BOTOX; Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo will be injected into the Glabellar Complex on Day 1.
  Interventions: Drug: Placebo
- OnabotulinumtoxinA X Dose A (Experimental): OnabotulinumtoxinA X Dose A will be injected into the Glabellar Complex on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X
- OnabotulinumtoxinA X Dose B (Experimental): OnabotulinumtoxinA X Dose B will be injected into the Glabellar Complex on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X
- OnabotulinumtoxinA X Dose C (Experimental): OnabotulinumtoxinA X Dose C will be injected into the Glabellar Complex on Day 1.
  Interventions: Drug: OnabotulinumtoxinA X

INTERVENTIONS:
Drug: OnabotulinumtoxinA X — Injection
  Arms: OnabotulinumtoxinA X Dose A; OnabotulinumtoxinA X Dose B; OnabotulinumtoxinA X Dose C
Drug: Placebo — Injection
  Arms: Placebo

SUMMARY:
This is a Phase 2, dose ranging study to evaluate the safety of OnabotulinumtoxinA X and to compare the efficacy of OnabotulinumtoxinA X and placebo for the treatment of Glabellar Lines in adult participants with moderate to severe GL.

ELIGIBILITY:
Inclusion Criteria:

* Participant has sufficient visual acuity without the use of eyeglasses (contact lens use is acceptable) to accurately assess their facial lines, in the opinion of the investigator.
* Participant has moderate or severe GL at maximum frown.

Exclusion Criteria:

* History of known immunization to any botulinum toxin serotype.
* History of known hypersensitivity to any botulinum toxin serotype, or any other constituents of the study drug or its excipients, and/or other products in the same class.
* Presence or history of any medical condition that may place the participant at increased risk following exposure to OnabotulinumtoxinA X or interfere with the study evaluation, including:
* Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.
* Facial nerve palsy.
* Infection or dermatological condition at the site of study drug injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (18):
- United States (18):
  - Advanced Research Associates - Glendale /ID# 230418, Glendale, Arizona
  - Westside Aesthetics /ID# 230305, Los Angeles, California
  - The Eye Research Foundation /ID# 232544, Newport Beach, California
  - The Research Center at The Maas Clinic /ID# 230685, San Francisco, California
  - Center for Dermatology and Dermatologic Surgery /ID# 230684, Washington D.C., District of Columbia
  - Steven Fagien MD Aesthetic Eyelid Plastic Surgery /ID# 232542, Boca Raton, Florida
  - Baumann Cosmetic and Research Institute /ID# 232545, Miami, Florida
  - Research Institute of the Southeast, LLC /ID# 230436, West Palm Beach, Florida
  - Coleman Center For Cosmetic Dermatologic Surgery /ID# 230693, Metairie, Louisiana
  - Etre Cosmetic Dermatology and Laser Center /ID# 230437, New Orleans, Louisiana
  - SLUCare Cosmetic Dermatology /ID# 230333, St Louis, Missouri
  - Laser & Skin Surgery Center of New York /ID# 230683, New York, New York
  - Skin Search of Rochester Inc. /ID# 242540, Rochester, New York
  - Aesthetic Solutions /ID# 230716, Chapel Hill, North Carolina
  - Wilmington Dermatology Center /ID# 242544, Wilmington, North Carolina
  - Aventiv Research Dublin /ID# 232546, Dublin, Ohio
  - Westlake Dermatology & Cosmetic Surgery - Westlake /ID# 232543, Austin, Texas
  - Premier Clinical Research /ID# 230682, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Started | 45 | 90 | 92 | 101
Completed | 37 | 79 | 79 | 87
Not Completed | 8 | 11 | 13 | 14
Not completed — Lost to Follow-up | 5 | 8 | 3 | 6
Not completed — Withdrawal by Subject | 3 | 3 | 9 | 7
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Placebo: Placebo was injected into the Glabellar Complex on Day 1.
- OnabotulinumtoxinA X Dose A: OnabotulinumtoxinA X Dose A was injected into the Glabellar Complex on Day 1.
- OnabotulinumtoxinA X Dose B: OnabotulinumtoxinA X Dose B was injected into the Glabellar Complex on Day 1.
- OnabotulinumtoxinA X Dose C: OnabotulinumtoxinA X Dose C was injected into the Glabellar Complex on Day 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C | Total
Number analyzed (Participants) | 45 | 90 | 92 | 101 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.16) | 49.3 (12.19) | 46.9 (11.35) | 50.4 (13.34) | 48.8 (12.35)
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 1 | 1 | 1 | 3 | 6
  26-40 years | 9 | 21 | 30 | 19 | 79
  41-55 years | 25 | 42 | 43 | 43 | 153
  56-64 years | 6 | 12 | 11 | 21 | 50
  ≥65 years | 4 | 14 | 7 | 15 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 77 | 75 | 90 | 282
  Male | 5 | 13 | 17 | 11 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 17 | 15 | 15 | 58
  Not Hispanic or Latino | 34 | 73 | 77 | 86 | 270
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 7 | 2 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 6 | 3 | 8 | 19
  White | 41 | 77 | 84 | 88 | 290
  More than one race | 0 | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Achievement of ≥ 1-grade Improvement From Baseline as Rated by Investigator Using the Clinician Glabellar Lines Scale.
Description: The Clinician Glabellar Lines Scale is a four point scale used to assess the severity of Glabellar Lines at maximum contraction ranging from 0 - None to 3 - Severe
Time Frame: Day 1 to Day 30
Population: Multiple Imputation - Intent-to-Treat Population
  Estimated responder is the average number of responders across 5 imputed datasets.
  Confidence interval for responder rate is calculated using normal approximation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 45 | 90 | 92 | 101
percentage of participants | 17.8 [6.6 to 28.9] | 95.6 [91.3 to 99.8] | 98.9 [96.8 to 100.0] | 98.0 [95.3 to 100.0]

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: Day 1 to Day 270
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 45 | 90 | 91 | 99
Participants
  Treatment-Emergent Adverse Events (TEAE) | 23 | 34 | 30 | 44
  TEAE Related to Study Treatment | 7 | 13 | 10 | 15
  TEAE Related to Study Procedure | 7 | 10 | 10 | 14
  TEAE Related to Study Drug | 7 | 13 | 10 | 15

3. Secondary Outcome: Percentage of Participants With Achievement of None or Mild as Rated by Investigator Using the Clinician Glabellar Lines Scale.
Description: as for outcome 1
Time Frame: Day 1 to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 45 | 90 | 92 | 101
percentage of participants | 6.7 [0.0 to 14.0] | 90.0 [83.8 to 96.2] | 93.5 [88.4 to 98.5] | 95.0 [90.8 to 99.3]

4. Secondary Outcome: Percentage of Participants With Achievement of Improvement Per the Facial Lines Satisfaction Questionnaire Impact Domain, Among Subjects With Baseline Scores of 14 Points or Greater.
Description: The Facial Line Satisfaction Questionnaire assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the subject perspective.
  Domain scores are calculated as the mean of transformed item scores on a 0 (low impact) to 100 (highest negative impact) scale.
Time Frame: Day 1 to Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 45 | 90 | 92 | 101
percentage of participants | 42.2 [27.8 to 56.7] | 65.6 [55.7 to 75.4] | 71.7 [62.5 to 80.9] | 73.3 [64.6 to 81.9]

5. Secondary Outcome: Percentage of Participants With Achievement of Satisfaction With Treatment Per the Facial Line Satisfaction Questionnaire Item 5.
Description: The Facial Line Satisfaction Questionnaire assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the subject perspective.
  A score of 100 represents the best score (very satisfied) and a score of 0 represent the worst score (very dissatisfied) on the satisfaction domain or satisfaction single items.
Time Frame: Day 1 to Day 60
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
Number analyzed (Participants) | 45 | 90 | 92 | 101
percentage of participants | 4.4 [0.0 to 10.5] | 80.0 [71.7 to 88.3] | 78.3 [69.8 to 86.7] | 87.1 [80.6 to 93.7]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 268, 267, 269, and 269 days for Placebo, OnabotulinumtoxinA X Dose A, Dose B and Dose C, respectively.
Arm/Group | Placebo | OnabotulinumtoxinA X Dose A | OnabotulinumtoxinA X Dose B | OnabotulinumtoxinA X Dose C
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/90 | 0/91 | 0/99
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/90 | 0/91 | 2/99
Other Adverse Events (participants affected / at risk) | 11/45 | 15/90 | 14/91 | 22/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | OnabotulinumtoxinA X Dose A (N=90) | OnabotulinumtoxinA X Dose B (N=91) | OnabotulinumtoxinA X Dose C (N=99)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMNIOTIC CAVITY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | OnabotulinumtoxinA X Dose A (N=90) | OnabotulinumtoxinA X Dose B (N=91) | OnabotulinumtoxinA X Dose C (N=99)
EYELID PTOSIS (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 8 (8)
INJECTION SITE OEDEMA (General disorders) | 1 (1) | 5 (5) | 2 (2) | 4 (4)
INJECTION SITE PAIN (General disorders) | 4 (5) | 4 (4) | 5 (5) | 5 (5)
COVID-19 (Infections and infestations) | 8 (8) | 9 (9) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT05100199/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT05100199/SAP_001.pdf